CLINICAL TRIAL: NCT05607056
Title: Phase 4, Efficacy and Safety of Sinquanon for Prevention of Antibiotic-associated Diarrhea in Adults in the Out-patient Setting: Prospective, Multicenter, Double-blind, Placebo-controlled Randomized Parallel-arm Clinical Study
Brief Title: Efficacy and Safety of Sinquanon for Prevention of Antibiotic-associated Diarrhea in Adults
Acronym: SPAADA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neopharm Bulgaria Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SPAADA202211_001; 2022-002817-40 (EudraCT Number)
Record Dates: First submitted 2022-10-31; First posted 2022-11-07 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2022-12

CONDITIONS: Antibiotic-associated Diarrhea
Keywords: Probiotics; Antibiotics; Antibiotic-associated diarrhea; High-dose; Multistrain

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, double-blind, placebo-controlled, randomized, parallel-arm clinical study
Who Masked: Participant, Investigator
Masking Description: Investigators will be provided with coded and identical products. Each individual involved in the study will be blinded to the assignment until study completion. Considering the established safety profile of the probiotic strains no necessity is foreseen for urgent unblinding of treatment assignment. With this in mind, no copies of the treatment assignments will be stored at the enrollment sites. If needed, the Investigators may receive information about the assignment of a particular subject only after review and approval by the Medical monitor. No information about the subjects will be shared with the company conducting the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): During the antibiotic dosing (from 5 to 10 days): 2 capsules once a day 2 hours before or 2 hours after antibiotic administration. 14 days following completion of antibiotic dosing: 1 capsule a day.
  Interventions: Dietary Supplement: Sinquanon
- Placebo (Placebo Comparator): During the antibiotic dosing (from 5 to 10 days): 2 capsules once a day 2 hours before or 2 hours after antibiotic administration. 14 days following completion of antibiotic dosing: 1 capsule a day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Sinquanon — This probiotic food supplement includes fourteen probiotic bacterial strains of Lactobacillus Spp, Bifidobacterium Spp., Bacillus coagulans, Saccharomyces boulardii, three prebiotics and Vitamin-B complex - B1, B2, B3, B6, B7, B9 in an enterosolvent cellulose capsule. The product includes supplementary substances: maltodextrin and magnesium stearate.
  2 capsules once a day during the antibiotic dosing. 1 capsule a day for 14 days following completion of antibiotic dosing.
  Arms: Probiotic
Dietary Supplement: Placebo — The placebo product will have the same appearance as the active product and the same composition but without the live bacteria, prebiotics, and vitamin-B complex. 2 capsules once a day during the antibiotic dosing. 1 capsule a day for 14 days following completion of antibiotic dosing.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of a probiotic, SINQUANON, on the reduction of the occurrence of diarrhea associated with antibiotic use in adults.

DETAILED DESCRIPTION:
The study aims to evaluate the efficacy of a specialized multi-strain probiotic, SINQUANON, on the reduction of the incidence of antibiotic-associated diarrhea in adults and to demonstrate the benefit of administering the specialized multi-strain probiotic as a routine add-on to antibiotic therapy on prevention of antibiotic-associated diarrhea in adults who take antibiotics in the outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged 18 to 60 years.
* The subject has given written informed consent after being provided orally with information about the study objective and design, including the administration regimen of the studied probiotic and the study procedures, the available safety data, as well as the rights and obligations of a participant.
* The subject initiates oral antibiotic treatment in the ambulatory setting.
* Acceptable antibiotic therapy:

  * Broad-spectrum penicillins
  * Cephalosporins
  * Quinolones
  * Tetracyclines

Sequential administration of two antibiotics from the allowed groups is permitted, if the total duration of the antibiotic treatment does not exceed 10 days.

* Planned duration of the antibiotic treatment of 5 to 10 days.
* Body mass index (BMI) of 18.0 to 29.9 kg/m2
* In the opinion of the Investigator, the subject can adhere to the visit schedule, to be compliant with the trial treatment regimen and to complete the study.
* The patient has a smartphone and can use it.

Exclusion Criteria:

* Antibiotics use within 60 days prior to randomization.
* Daily consumption of probiotics, yogurt with probiotics and inability to stop this consumption.
* Use of antidiarrheal medications, laxatives, enemas, or suppositories within 1 week prior to randomization and for the duration of the trial.
* An episode of diarrhea within 30 days before screening, defined as ≥3 loose or liquid stools over 24 hours, regardless of the cause of the diarrhea.
* Acute or chronic constipation - average number of formed stools <3 per week.
* Allergy or hypersensitivity to any of the ingredients of the trial product.
* Allergy or hypersensitivity to the antibiotic prescribed on Day 1.
* Prior documented infection with Clostridioides difficile ≤3 months before screening.
* History of chronic gastrointestinal conditions, including irritable bowel syndrome, chronic constipation, chronic diarrhea, dyspepsia, gastroesophageal reflux disease, diverticulitis, ulcerative colitis, Crohn's disease or any other abnormality in the absorption or gastrointestinal dysfunction.
* Use of proton-pump inhibitors (PPIs) within 30 days prior to Day 1 and for the duration of the study.
* Surgery to the intestines, artificial heart valve, history of rheumatological heart disease or infectious endocarditis within one year prior to screening.
* Immunosuppressive therapy or any condition causing immunosuppression (including hematologic malignancies, AIDS, long-lasting corticosteroid treatment).
* Planned administration of antibiotics, different from those acceptable for the study.
* Patients in severe condition requiring urgent hospitalization or planned hospitalization during the study.
* Planned administration of antibiotics >10 days.
* BMI ≥ 30 kg/m2.
* Pregnant or lactating women; women who plan to get pregnant during the study.
* Drug abuse or alcohol within the past year.
* Unstable medical conditions, in the judgement of the Investigator.
* Eating disorders (for example, anorexia, bulimia).
* On a vegan diet.
* Participation in a clinical trial within 60 days prior to randomization.
* Inability to comply with the study protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 565 (Actual)
Dates: Start 2022-11-27 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Incidence of Antibiotic-Associated diarrhea (AAD) | By 21+2 days after completion of antibiotic dosing.
  The incidence of AAD is defined as the number of subjects who experience at least one day of diarrhea compared to the total number of subjects enrolled in the given treatment arm. AAD is defined as 3 or more loose or liquid stools (types 5-7 according to Bristol Stool Scale [BSS]) over a period of 24 hours.

SECONDARY OUTCOMES:
Severity of AAD | By 21+2 days after completion of antibiotic dosing.
  Investigator will assess AAD severity using the following modified scale defining AAD as: severe: ≥7 unformed/loose/liquid stools; moderate: 5-6 unformed/loose/liquid stools; mild: a change in the stool pattern 3-4 unformed/loose/liquid stools a day. Investigator's assessment will take into consideration the 24-hour period presenting with the worst severity.
Duration of diarrhea | By 21+2 days after completion of antibiotic dosing.
  Number of sequential days with diarrhea. Defined as the time until the first normalization of the stool form according to BSS: presence of one or two sequential normal stools, i.e. "soft and formed" or "hard and formed" - types 1-4 per BSS (or lack of stool) for a period of 24 hours.
Antibiotic-associated adverse experiences (abdominal pain, bloating, passing gas, nausea) | By 21+2 days after completion of antibiotic dosing.
  Presence of abdominal pain, bloating, passing gass, nausea - Yes/No.
Visual-analogue scale for the gastrointestinal quality of life (VAS-QoL) | By 21+2 days after completion of antibiotic dosing.
  Measured via Visual-analogue scale for the gastrointestinal quality of life. The subjects will answer the question: "To what extent the abdominal problems impact your quality of life?" This scale has numerical points from 0 to 100. "100" indicates THE WORST quality of life one can imagine, "0" indicates NO problems and THE BEST quality of life one can imagine.
Adverse events (AE) | By 21+2 days after completion of antibiotic dosing.
  Incidence of mild (for example, self-resolving), moderate (for example, those requiring medical evaluation) and serious AEs (for example, events requiring lasting hospitalization) adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Georgi Momekov, Prof PhD, Principal Investigator — Department of Pharmacology, Pharmacotherapy and Toxicology, Medical University of Sofia; Karen Dzhambazov, Prof, PhD, Principal Investigator — University hospital for active treatment Sveti Georgi, Medical University-Plovdiv; Nikolay Sapundziev, Prof, PhD, Principal Investigator — Department of Neurosurgery and Otorhinolaryngology, Medical University - Varna; Milena Encheva, MD, PhD, Principal Investigator — Military Medical Academy, Bulgaria; Boris Bogov, Prof, PhD, Principal Investigator — UMHAT "Sveta Anna"; Rosen Nikolov, Prof, MD, Principal Investigator — UMHAT St Ivan Rilski; Rumen Benchev, Prof, Principal Investigator — Hill Clinic; Vladimir Hodzhev, Prof, PhD, Principal Investigator — University Hospital "St George"; Spiridon Todorov, Prof, PhD, Principal Investigator — University Hospital "Tsaritsa Yoanna - ISUL"; Vania Youroukova, Prof, PhD, Principal Investigator — University Hospital for Pulmonary Diseases " St. Sofia"
Locations (3):
- Bulgaria (3):
  - University Hospital "St George", Plovdiv
  - University Hospital for Pulmonary Diseases " St. Sofia", Sofia
  - University Hospital "Tsaritsa Yoanna - ISUL", Sofia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Konstantinidis T, Tsigalou C, Karvelas A, Stavropoulou E, Voidarou C, Bezirtzoglou E. Effects of Antibiotics upon the Gut Microbiome: A Review of the Literature. Biomedicines. 2020 Nov 16;8(11):502. doi: 10.3390/biomedicines8110502. PMID 33207631
- [Background] Francino MP. Antibiotics and the Human Gut Microbiome: Dysbioses and Accumulation of Resistances. Front Microbiol. 2016 Jan 12;6:1543. doi: 10.3389/fmicb.2015.01543. eCollection 2015. PMID 26793178
- [Background] Mekonnen SA, Merenstein D, Fraser CM, Marco ML. Molecular mechanisms of probiotic prevention of antibiotic-associated diarrhea. Curr Opin Biotechnol. 2020 Feb;61:226-234. doi: 10.1016/j.copbio.2020.01.005. Epub 2020 Feb 19. PMID 32087535
- [Background] Barbut F, Meynard JL. Managing antibiotic associated diarrhoea. BMJ. 2002 Jun 8;324(7350):1345-6. doi: 10.1136/bmj.324.7350.1345. No abstract available. PMID 12052785
- [Background] Szajewska H, Kolodziej M. Systematic review with meta-analysis: Lactobacillus rhamnosus GG in the prevention of antibiotic-associated diarrhoea in children and adults. Aliment Pharmacol Ther. 2015 Nov;42(10):1149-57. doi: 10.1111/apt.13404. Epub 2015 Sep 13. PMID 26365389
- [Background] Szajewska H, Kolodziej M. Systematic review with meta-analysis: Saccharomyces boulardii in the prevention of antibiotic-associated diarrhoea. Aliment Pharmacol Ther. 2015 Oct;42(7):793-801. doi: 10.1111/apt.13344. Epub 2015 Jul 27. PMID 26216624
- [Background] Ouwehand AC. A review of dose-responses of probiotics in human studies. Benef Microbes. 2017 Apr 26;8(2):143-151. doi: 10.3920/BM2016.0140. Epub 2016 Dec 23. PMID 28008787
- [Background] Szajewska H, Canani RB, Guarino A, Hojsak I, Indrio F, Kolacek S, Orel R, Shamir R, Vandenplas Y, van Goudoever JB, Weizman Z; ESPGHAN Working Group for ProbioticsPrebiotics. Probiotics for the Prevention of Antibiotic-Associated Diarrhea in Children. J Pediatr Gastroenterol Nutr. 2016 Mar;62(3):495-506. doi: 10.1097/MPG.0000000000001081. PMID 26756877
- [Background] Goldenberg JZ, Lytvyn L, Steurich J, Parkin P, Mahant S, Johnston BC. Probiotics for the prevention of pediatric antibiotic-associated diarrhea. Cochrane Database Syst Rev. 2015 Dec 22;(12):CD004827. doi: 10.1002/14651858.CD004827.pub4. PMID 26695080
- [Background] Gao XW, Mubasher M, Fang CY, Reifer C, Miller LE. Dose-response efficacy of a proprietary probiotic formula of Lactobacillus acidophilus CL1285 and Lactobacillus casei LBC80R for antibiotic-associated diarrhea and Clostridium difficile-associated diarrhea prophylaxis in adult patients. Am J Gastroenterol. 2010 Jul;105(7):1636-41. doi: 10.1038/ajg.2010.11. Epub 2010 Feb 9. PMID 20145608
- [Derived] Hodzhev V, Dzhambazov K, Sapundziev N, Encheva M, Todorov S, Youroukova V, Benchev R, Nikolov R, Bogov B, Momekov G, Hadjiev V. High-dose Probiotic Mix of Lactobacillus spp., Bifidobacterium spp., Bacillus coagulans, and Saccharomyces boulardii to Prevent Antibiotic-associated Diarrhea in Adults: A Multicenter, Randomized, Double-blind, Placebo-controlled Trial (SPAADA). Open Forum Infect Dis. 2024 Oct 21;11(11):ofae615. doi: 10.1093/ofid/ofae615. eCollection 2024 Nov. PMID 39529939